CLINICAL TRIAL: NCT02905266
Title: Phase IIIb, Randomized, Study of Multiple Administration Regimens for Nivolumab Plus Ipilimumab in Subjects With Previously Untreated Unresectable or Metastatic Melanoma
Brief Title: A Safety and Efficacy Study of Multiple Administration Regimens for Nivolumab Plus Ipilimumab in Subjects With Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-742; 2016-001941-26 (EudraCT Number)
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nivolumab and Ipilimumab Concomitant Administration (Experimental): Followed by Nivolumab monotherapy
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Nivolumab and Ipilimumab Sequential Administration (Experimental): Followed by Nivolumab monotherapy
  Interventions: Biological: Nivolumab; Biological: Ipilimumab

INTERVENTIONS:
Biological: Nivolumab — -Specified dose on specified days
Biological: Ipilimumab — -Specified dose on specified days

SUMMARY:
This is a safety and efficacy study of different administration regimens of nivolumab plus Ipilimumab in subjects with previously untreated, unresectable or metastatic melanoma.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Males and Females, ages 15 years ≥ of age (Except where local regulations and/or institutional policies do not allow for subjects < 18 years of age to participate)
* Subjects must have been diagnosed with stage III or/and stage IV histologically confirmed melanoma that is unresectable or metastatic
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Subjects have not been treated by systemic anticancer therapy for unresectable or metastatic melanoma

Exclusion Criteria:

* Subjects with active brain metastases or leptomeningeal metastases
* Subjects with ocular melanoma
* Subjects with active, known or suspected autoimmune disease

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2019-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (16):
- Australia (3):
  - Melanoma Institute Australia, North Sydney, New South Wales
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Cabrini Hospital, Malvern, Victoria
- France (6):
  - Local Institution, Lyon
  - Hopital De La Timone, Marseille
  - Local Institution, Nantes
  - Hopital Saint Louis, Paris
  - Local Institution, Paris
  - Hopital Trousseau - Chru Tours, Tours
- Italy (4):
  - Istituto Nazionale Per La Ricerca Sul Cancro - Oncologia Med, Genova
  - Istituto Scientifico Romagnolo Per Lo Studio E Cura Tumori, Meldola (FC)
  - Istituto Europeo Di Oncologia, Milan
  - Azienda Ospedaliera Citta della Salute e della Scienza, Torino
- Spain (3):
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Seville

REFERENCES:
- [Derived] Menzies AM, Salman P, Frontera OA, Pook D, Hocking CM, Zakharia Y, Gurney H, Gedye C, Goh JC, Telivala B, Grob JJ, Lebbe C, de la Cruz Merino L, Machet L, Neidhardt EM, Qureshi A, Hosein F, Hamuro L, Simsek B, Amin A. Administration of nivolumab plus ipilimumab: Infusion of the fixed-ratio combination versus sequential infusions in two randomized controlled trials of metastatic melanoma (CheckMate 742) and renal cell carcinoma (CheckMate 800). Cancer. 2025 Jul 15;131(14):e35962. doi: 10.1002/cncr.35962. PMID 40614118
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 106 participants were randomized and treated.
Groups:
- Fixed Ratio Combination: Concomitant administration of Nivolumab and Ipilimumab (1:3 protein-mass ratio) every 3 weeks for 4 doses followed by Nivolumab flat dose in the Maintenance Phase
- Sequential Combination: Sequential administration of Nivolumab and Ipilimumab every 3 weeks for 4 doses followed by Nivolumab flat dose in the Maintenance Phase
Period: Treatment Phase Part 1
Arm/Group | Fixed Ratio Combination | Sequential Combination
Started (Randomized and treated) | 53 | 53
Completed (Completed = Continuing in study) | 24 | 30
Not Completed | 29 | 23
Not completed — Participant Withdrew Consent | 1 | 0
Not completed — Disease Progression | 6 | 7
Not completed — Study Drug Toxicity | 22 | 16
Period: Transition From Part 1 to Part 2
Arm/Group | Fixed Ratio Combination | Sequential Combination
Started | 24 | 30
Completed | 20 | 22
Not Completed | 4 | 8
Not completed — Adverse event unrelated to study drug | 1 | 0
Not completed — Disease progression | 2 | 1
Not completed — Study drug toxicity | 0 | 4
Not completed — Death | 0 | 1
Not completed — Participant withdrew consent | 0 | 1
Not completed — Adverse Event | 1 | 1
Period: Maintenance Phase Part 2
Arm/Group | Fixed Ratio Combination | Sequential Combination
Started | 20 | 22
Completed | 8 | 14
Not Completed | 12 | 8
Not completed — Disease Progression | 9 | 2
Not completed — Study Drug Toxicity | 3 | 4
Not completed — Maximum Clinical Benefit | 0 | 2

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Fixed Ratio Combination | Sequential Combination | Total
Number analyzed (Participants) | 53 | 53 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (14.5) | 56.3 (14.6) | 57.2 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 26 | 44
  Male | 35 | 27 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 26 | 28 | 54
  Unknown or Not Reported | 26 | 24 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 48 | 50 | 98
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants Affected by AEs in the Narrow Scope MedDRA Anaphylactic Reaction SMQ
Description: This outcome describes the percentage of participants experiencing at least 1 AE in the MedDRA Anaphylactic Reaction narrow scope SMQ. The narrow scope SMQ is composed of a large list of terms, including (but not limited to) anaphylactic shock and reaction, shock and shock symptoms, and circulatory collapse, among the others.
Time Frame: Within 2 days from administration of any of the 4 doses in part 1 period (approximately 12 weeks)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Fixed Ratio Combination | Sequential Combination
Number analyzed (Participants) | 53 | 53
Percent of Participants | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 6.7]
Statistical Analysis 1: Comparison: Fixed Ratio Combination vs Sequential Combination; Test type: Superiority; Percent Difference in incidence rates = 0.0, 95% CI 2-sided [0.0 to 0.0] — Fixed Ratio Combination over Sequential Combination

2. Secondary Outcome: Percentage of Participants Affected by Hypersensitivity/Infusion Reaction Select AEs
Description: This outcome describes the percentage of participants experiencing at least 1 AE in the Hypersensitivity/Infusion select AEs category. The select AEs consist of a list of preferred terms defined by the Sponsor and represent AEs with a potential immune-mediated etiology. The following 5 MedDRA preferred terms are included in the hypersensitivity/infusion reaction select AE category: Anaphylactic Reaction, Anaphylactic Shock, Bronchospasm, Hypersensitivity, and Infusion Related Reaction
Time Frame: Within 2 days from administration of any of the 4 doses in part 1 period (approximately 12 weeks)
Population: All treated participants
Measure: Number; unit: Percent of Participants
Arm/Group | Fixed Ratio Combination | Sequential Combination
Number analyzed (Participants) | 53 | 53
Percent of Participants | 7.5 | 9.4

3. Secondary Outcome: Percentage of Participants Affected by All Causality Grade 3 - 5 AEs
Description: This outcome describes the percentage of participants who experienced at least 1 AE of Grade 3 or higher defined using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 criteria
Time Frame: From initial dose of study treatment and within 30 days of the last dose of study treatment (approximately 25 months)
Population: All treated participants
Measure: Number; unit: Percent of participants
Arm/Group | Fixed Ratio Combination | Sequential Combination
Number analyzed (Participants) | 53 | 53
Percent of participants | 69.8 | 56.6

4. Secondary Outcome: Percentage of Participants Affected by Drug-related Grade 3 - 5 AEs
Description: This outcome describes the percentage of participants who experienced at least 1 Drug-related AE of Grade 3 or higher defined using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 criteria
Time Frame: From initial dose of study treatment and within 30 days of the last dose of study treatment (approximately 25 months)
Population: All treated participants
Measure: Number; unit: Percent of participants
Arm/Group | Fixed Ratio Combination | Sequential Combination
Number analyzed (Participants) | 53 | 53
Percent of participants | 58.5 | 47.2

5. Secondary Outcome: Geometric Mean Concentration of Ipilimumab at End of Infusion (EOI)
Time Frame: From Cycle 1, Day 1 to Cycle 4, Day 1 (approximately 9 weeks). Each cycle lasts 3 weeks. Cycle 1 day 1, Cycle 2 day 1 and Cycle 4 day 1 values reported.
Population: All treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (ug/mL)
Arm/Group | Fixed Ratio Combination | Sequential Combination
Number analyzed (Participants) | 53 | 53
micrograms per milliliter (ug/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 48 | 49
  Cycle 1 Day 1 | 60.4 (93.0) | 61.5 (72.3)
  Cycle 2 Day 1: number analyzed (Participants) | 48 | 46
  Cycle 2 Day 1 | 66.8 (134) | 72.1 (71.8)
  Cycle 4 Day 1: number analyzed (Participants) | 22 | 30
  Cycle 4 Day 1 | 77.9 (94.2) | 84.6 (104)

6. Secondary Outcome: Geometric Mean Concentration of Nivolumab at End of Infusion (EOI)
Time Frame: as for outcome 5
Population: All treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (ug/mL)
Arm/Group | Fixed Ratio Combination | Sequential Combination
Number analyzed (Participants) | 53 | 53
micrograms per milliliter (ug/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 50 | 50
  Cycle 1 Day 1 | 20.9 (77.3) | 21.8 (117)
  Cycle 2 Day 1: number analyzed (Participants) | 48 | 46
  Cycle 2 Day 1 | 24.2 (122) | 22.4 (101)
  Cycle 4 Day 1: number analyzed (Participants) | 22 | 30
  Cycle 4 Day 1 | 27.9 (79.8) | 27.4 (79.9)

7. Secondary Outcome: Geometric Mean Trough Concentration of Ipilimumab
Time Frame: From Cycle 2, Day 1 to Cycle 4, Day 1 (approximately 6 weeks). Each cycle lasts 3 weeks.
Population: All treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (ug/mL)
Arm/Group | Fixed Ratio Combination | Sequential Combination
Number analyzed (Participants) | 53 | 53
micrograms per milliliter (ug/mL)
  Cycle 2 Day 1: number analyzed (Participants) | 45 | 49
  Cycle 2 Day 1 | 10.8 (30.2) | 9.94 (38.9)
  Cycle 4 Day 1: number analyzed (Participants) | 21 | 29
  Cycle 4 Day 1 | 16.5 (36.9) | 13.7 (46.0)

8. Secondary Outcome: Geometric Mean Trough Concentration of Nivolumab
Time Frame: From Cycle 2, Day 1 to Cycle 4, Day 1 (approximately 6 weeks). Each cycle lasts 3 weeks.
Population: All treated participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (ug/mL)
Arm/Group | Fixed Ratio Combination | Sequential Combination
Number analyzed (Participants) | 53 | 53
micrograms per milliliter (ug/mL)
  Cycle 2 Day 1: number analyzed (Participants) | 46 | 48
  Cycle 2 Day 1 | 3.94 (56.6) | 2.75 (65.9)
  Cycle 4 Day 1: number analyzed (Participants) | 19 | 27
  Cycle 4 Day 1 | 6.50 (44.6) | 4.05 (75.3)

9. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR is defined as the proportion of participants with a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR). The BOR is defined as the best response designation, as determined by the investigator, recorded between the date of randomization and the date of objectively documented progression per RECIST 1.1 or the date of subsequent anti-cancer therapy, whichever occurs first.
Time Frame: Week 12 following randomization, every 8 weeks for the first 12 months and then every 12 weeks until disease progression (approximately 20 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Fixed Ratio Combination | Sequential Combination
Number analyzed (Participants) | 53 | 53
Percentage of Participants | 52.8 [38.6 to 66.7] | 60.4 [46.0 to 73.5]
Statistical Analysis 1: Comparison: Fixed Ratio Combination vs Sequential Combination; Test type: Superiority; Percent Difference of ORRs = -7.5, 95% CI 2-sided [-26.1 to 11.0] — Cochran-Mantel-Haenszel (CMH) method of weighting
Statistical Analysis 2: Comparison: Fixed Ratio Combination vs Sequential Combination; Test type: Superiority; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.35 to 1.58]

10. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time between the date of randomization and the first date of documented progression, as determined by the investigator, or death due to any cause, whichever occurs first.
Time Frame: From the date of randomization to the first date of documented progression (approximately 26 months)
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Fixed Ratio Combination | Sequential Combination
Number analyzed (Participants) | 53 | 53
Months | 10.25 [2.96 to NA] — Upper limit not reached because of insufficient number of participants with an event | NA [4.96 to NA] — (Value) N.A.explanation: Below the level of detection (Upper limit) n/a explanation: Upper limit not reached because of insufficient number of participants with an event
Statistical Analysis 1: Comparison: Fixed Ratio Combination vs Sequential Combination; Test type: Superiority; Hazard Ratio (HR) = 1.36, 95% CI 2-sided [0.78 to 2.37] — Stratified Cox proportional hazard model

11. Primary Outcome: Percentage of Participants Affected by Adverse Events (AEs) in the Broad Scope MedDRA Anaphylactic Reaction Standardized MedDRA Queries (SMQ)
Description: This outcome describes the percentage of participants experiencing at least 1 AE in the MedDRA Anaphylactic Reaction broad scope SMQ. Such AEs include any acute systemic reaction characterized by a large list of terms, including (but not limited to) pruritus, urticaria, flushing, hypotension, respiratory distress, and vascular insufficiency. It also includes other signs and symptoms such as asthma, choking sensation, coughing, sneezing, and difficulty breathing due to laryngeal spasm and/or bronchospasm. Less frequent clinical presentations are also captured and include hyperventilation, sensation of foreign body, and ocular edema.
Time Frame: Within 2 days from administration of any of the 4 doses in part 1 period (approximately 12 weeks)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Fixed Ratio Combination | Sequential Combination
Number analyzed (Participants) | 53 | 53
Percent of Participants | 15.1 [6.7 to 27.6] | 17.0 [8.1 to 29.8]
Statistical Analysis 1: Comparison: Fixed Ratio Combination vs Sequential Combination; Test type: Superiority; Cochran-Mantel-Haenszel Odds Ratio = 0.87, 95% CI 2-sided [0.30 to 2.49] — Fixed Ratio Combination over Sequential Combination
Statistical Analysis 2: Comparison: Fixed Ratio Combination vs Sequential Combination; Test type: Superiority; Percent difference in incidence rates = -1.9, 95% CI 2-sided [-16.0 to 12.2] — Fixed Ratio Combination over Sequential Combination

ADVERSE EVENTS:
Time Frame: From first dose to 100 days following administration of the last dose (approximately 27 months).
Arm/Group | Fixed Ratio Combination | Sequential Combination
All-Cause Mortality (participants affected / at risk) | 14/53 | 14/53
Serious Adverse Events (participants affected / at risk) | 35/53 | 35/53
Other Adverse Events (participants affected / at risk) | 51/53 | 51/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fixed Ratio Combination (N=53) | Sequential Combination (N=53)
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Hypophysitis (Endocrine disorders) | 1 | 1
Thyroiditis (Endocrine disorders) | 2 | 1
Iridocyclitis (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Autoimmune colitis (Gastrointestinal disorders) | 2 | 1
Colitis (Gastrointestinal disorders) | 4 | 4
Cyclic vomiting syndrome (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Erosive duodenitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 3 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 2
Melaena (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1
Adverse drug reaction (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 8 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 2 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 2 | 1
Hepatocellular injury (Hepatobiliary disorders) | 6 | 3
Hypertransaminasaemia (Hepatobiliary disorders) | 2 | 0
Autoimmune disorder (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Meningitis aseptic (Infections and infestations) | 0 | 2
Parotitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2
Liver function test abnormal (Investigations) | 1 | 0
Pancreatic enzymes increased (Investigations) | 1 | 0
Pneumocystis test positive (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 7
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Meningorrhagia (Nervous system disorders) | 1 | 0
Motor neurone disease (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fixed Ratio Combination (N=53) | Sequential Combination (N=53)
Anaemia (Blood and lymphatic system disorders) | 3 | 6
Hyperthyroidism (Endocrine disorders) | 8 | 6
Hypophysitis (Endocrine disorders) | 2 | 4
Hypothyroidism (Endocrine disorders) | 11 | 8
Thyroiditis (Endocrine disorders) | 2 | 3
Abdominal distension (Gastrointestinal disorders) | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 4
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3
Colitis (Gastrointestinal disorders) | 1 | 5
Constipation (Gastrointestinal disorders) | 9 | 7
Diarrhoea (Gastrointestinal disorders) | 16 | 25
Dry mouth (Gastrointestinal disorders) | 6 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 9 | 12
Vomiting (Gastrointestinal disorders) | 9 | 12
Asthenia (General disorders) | 17 | 20
Chills (General disorders) | 4 | 4
Fatigue (General disorders) | 10 | 9
Influenza like illness (General disorders) | 3 | 8
Oedema peripheral (General disorders) | 5 | 5
Pyrexia (General disorders) | 14 | 18
Hepatitis (Hepatobiliary disorders) | 4 | 2
Hepatocellular injury (Hepatobiliary disorders) | 7 | 3
Bronchitis (Infections and infestations) | 2 | 3
Nasopharyngitis (Infections and infestations) | 1 | 4
Oral herpes (Infections and infestations) | 0 | 3
Sinusitis (Infections and infestations) | 1 | 3
Urinary tract infection (Infections and infestations) | 3 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 4
Alanine aminotransferase increased (Investigations) | 8 | 7
Amylase increased (Investigations) | 5 | 3
Aspartate aminotransferase increased (Investigations) | 6 | 5
Blood lactate dehydrogenase increased (Investigations) | 5 | 4
Gamma-glutamyltransferase increased (Investigations) | 3 | 2
Lipase increased (Investigations) | 8 | 5
Decreased appetite (Metabolism and nutrition disorders) | 10 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 8
Dizziness (Nervous system disorders) | 2 | 4
Headache (Nervous system disorders) | 8 | 15
Paraesthesia (Nervous system disorders) | 2 | 5
Insomnia (Psychiatric disorders) | 4 | 5
Sleep disorder (Psychiatric disorders) | 2 | 3
Dysuria (Renal and urinary disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Erythema (Skin and subcutaneous tissue disorders) | 3 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 3
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 17
Rash (Skin and subcutaneous tissue disorders) | 15 | 12
Rash pruritic (Skin and subcutaneous tissue disorders) | 9 | 7
Vitiligo (Skin and subcutaneous tissue disorders) | 9 | 5
Deep vein thrombosis (Vascular disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT02905266/Prot_002.pdf
  • Statistical Analysis Plan (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT02905266/SAP_003.pdf